CLINICAL TRIAL: NCT00243555
Title: Molecular Analysis of Immuno-Regulatory Genes Expressed by Mononuclear Cells From Peanut Skin Test Positive Individuals With and Without a History of Peanut Ingestion
Brief Title: Development of an Algorithm to Better Predict Clinical Responsiveness to Peanut
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Food Allergy Initiative (Other); AllerGen NCE Inc. (Industry)
Organization: McMaster University (Other)
Other Study IDs: 2002H05183; FP-2005-25
Record Dates: First submitted 2005-10-20; First posted 2005-10-24 (Estimated); Last update posted 2007-02-01 (Estimated); Status verified 2006-09

CONDITIONS: Peanut Hypersensitivity
Keywords: peanut hypersensitivity; chemokines; cytokines; RNA,messenger; monocytes
MeSH Terms: conditions — Peanut Hypersensitivity | interventions — Skin Tests; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: allergy skin testing
Procedure: venepuncture

SUMMARY:
The purpose of this study is to develop a tool to better predict clinical allergy to peanut, so that those who are skin test positive but non allergic will not have to unnecessarily avoid peanut, and those with true allergy can be diagnosed, possibly without oral ingestion challenge, and treated appropriately

DETAILED DESCRIPTION:
Peanut allergy occurs in about 1% of the population. Allergic reactions to peanuts and tree nuts account for the majority of fatal and near fatal food allergic reactions. Currently the only available treatment is complete avoidance of peanut. Despite avoidance, the majority of peanut allergic people will accidentally ingest peanut. Accurate diagnosis is critical, yet often problematic. Current diagnostic methods such as skin and blood tests cannot predict definitively who is allergic and can result in patients being falsely labeled. One such group is children who have never been exposed to peanut as a means of preventing allergy, yet have positive skin tests. The only means of definitively diagnosing this group is with an oral peanut challenge, a potentially risky procedure. Previous studies have demonstrated differences in certain genes and growth factors between peanut allergic and non-allergic individuals. The proposed study has 2 phases. The first phase, almost completed, examines expression of genes and growth factors in defined groups of peanut allergic and non-allergic individuals which should help distinguish between these groups. Peripheral blood mononuclear cells from each patient will be cultured and analyzed for a variety of growth factors and other immune molecules, including mRNA, thought to be important in allergy.

The second phase of this study will involve feeding peanut to individuals with positive skin tests, who have never been peanut exposed. Their blood will be examined before and after the challenge using information from Part 1, and results will be correlated with their ability to tolerate peanut on feeding. This study should enable us to better predict who is truly peanut allergic.

There are four groups of patients in this study. Group 1 consists of individuals who are allergic to peanut. This group of individuals will have a positive skin test to peanut and a previous allergi reaction to peanut. Group 2 consists of indivduals who have a positive skin test to peanut but who are able to ingest peanuts without problems. Group 3 consists of individuals who have a positive skin test to peanut but who have no known ingestion of peanut and who have avoided peanut lifelong for whatever reason (e.g. a strong family history of peanut allergy). Lastly, group 4 consists of control subjects who are negative to the peanut skin test and are able to tolerate peanut without problems.

ELIGIBILITY:
Inclusion Criteria:

* 5 years of age and older
* Informed consent (Subject has provided an appropriately signed and dated informed consent. An appropriately signed and dated assent must be obtained from the parents or guardian if the subject is a child under 18 years of age.)
* Free of any clinically significant disease, such as uncontrolled asthma, which may interfere with study evaluations

Group 1:

* skin test positive to peanut
* documented clinical history of peanut allergy. A documented clinical history may include symptoms such as hives,swelling of the mouth or tongue, throat closing sensation, shortness of breath, wheezing, lightheadedness, anaphylaxis.

Group 2:

* Positive skin test to peanut
* History of being able to tolerate peanut exposure without problems

Group 3:

* Positive skin test to peanut
* No known ingestion of peanut

Group 4:

* Negative skin test to peanut
* Negative skin test to other food and environmental allergens
* Able to tolerate peanut exposure without problems

Exclusion Criteria:

* Women who are pregnant or nursing
* use of antihistamines or decongestant therapy four days prior to clinic visit
* use of nasal or inhaled corticosteroid in the 1 month period prior to clinic visit
* use of non-steroidal anti-inflammatory drugs (NSAIDS) in the week prior to clinic visit
* Moderate or severe/ uncontrolled asthma (defined as the use of more than 4 puffs of ventolin per day, not including prophylactic medications prior to exercise)
* Symptomatic allergic rhinitis
* Patients who had an acute allergic reaction to food, drugs, and bee sting in the 1 month period prior to clinic visit
* Use of an epi-pen during the past month
* respiratory infection one month prior to clinic visit
* immunotherapy

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2002-09

CONTACTS AND LOCATIONS:
Overall Officials: Susan Waserman, MSc, MD, FRCPC, Principal Investigator — Hamilton Health Sciences Corporation, McMaster Site
Locations (1):
- Hamilton Health Sciences Corporation, McMaster Site, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Heaton T, Rowe J, Turner S, Aalberse RC, de Klerk N, Suriyaarachchi D, Serralha M, Holt BJ, Hollams E, Yerkovich S, Holt K, Sly PD, Goldblatt J, Le Souef P, Holt PG. An immunoepidemiological approach to asthma: identification of in-vitro T-cell response patterns associated with different wheezing phenotypes in children. Lancet. 2005 Jan 8-14;365(9454):142-9. doi: 10.1016/S0140-6736(05)17704-6. PMID 15639296
- [Background] Turcanu V, Maleki SJ, Lack G. Characterization of lymphocyte responses to peanuts in normal children, peanut-allergic children, and allergic children who acquired tolerance to peanuts. J Clin Invest. 2003 Apr;111(7):1065-72. doi: 10.1172/JCI16142. PMID 12671056
- [Background] Umetsu DT. Revising the immunological theories of asthma and allergy. Lancet. 2005 Jan 8-14;365(9454):98-100. doi: 10.1016/S0140-6736(05)17714-9. No abstract available. PMID 15639274
- [Background] Kagan RS, Joseph L, Dufresne C, Gray-Donald K, Turnbull E, Pierre YS, Clarke AE. Prevalence of peanut allergy in primary-school children in Montreal, Canada. J Allergy Clin Immunol. 2003 Dec;112(6):1223-8. doi: 10.1016/j.jaci.2003.09.026. PMID 14657887
- [Background] Sampson HA. Update on food allergy. J Allergy Clin Immunol. 2004 May;113(5):805-19; quiz 820. doi: 10.1016/j.jaci.2004.03.014. PMID 15131561
- [Background] Roberts G, Lack G. Diagnosing peanut allergy with skin prick and specific IgE testing. J Allergy Clin Immunol. 2005 Jun;115(6):1291-6. doi: 10.1016/j.jaci.2005.02.038. PMID 15940149
- [Background] van Odijk J, Ahlstedt S, Bengtsson U, Borres MP, Hulthen L. Double-blind placebo-controlled challenges for peanut allergy the efficiency of blinding procedures and the allergenic activity of peanut availability in the recipes. Allergy. 2005 May;60(5):602-5. doi: 10.1111/j.1398-9995.2005.00666.x. PMID 15813803